CLINICAL TRIAL: NCT07094581
Title: Evaluation of the Effect of Adenoid Hypertrophy on the Masseter Muscle in Children: A Comparative Ultrasonographic Study
Status: Recruiting | Type: Observational
Sponsor: Melis AKYILDIZ (Other)
Responsible Party: Sponsor-Investigator, Melis AKYILDIZ, Assistant Professor, Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Other Study IDs: 2023/37
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-07

CONDITIONS: Adenoid Hypertrophy; Masseter Muscle; Malocclusion
Keywords: Adenoid Hypertrophy; Ultrasonography; Masseter Muscle
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adenoid Hypertrophy Group: Children aged 3-8 years diagnosed with adenoid hypertrophy.
  Interventions: Diagnostic Test: USG
- Healthy Control Group: Healthy children aged 3-8 years without adenoid hypertrophy.
  Interventions: Diagnostic Test: USG

INTERVENTIONS:
Diagnostic Test: USG — Masseter Muscle Thickness and Internal Echogenic Bands Assessed by Ultrasonography

SUMMARY:
The goal of this observational study is to evaluate the effect of adenoid hypertrophy on the masseter muscle in children aged 3 to 8 years. The primary objectives are:

* To assess whether adenoid hypertrophy affects the thickness or structure of the masseter muscle.
* To determine whether there is a measurable difference in masseter muscle characteristics between children with and without adenoid hypertrophy.

Researchers will compare children diagnosed with adenoid hypertrophy and scheduled for adenoidectomy to healthy controls without adenoid hypertrophy.

Each participant will:

* Undergo ultrasonographic examination of the masseter muscle using a 9L linear probe (6-15 MHz), and
* Have their occlusal relationship, dental findings, age, sex, and adenoid hypertrophy grade recorded.

DETAILED DESCRIPTION:
Hypotheses

H0 (Null Hypothesis): There is no difference in masseter muscle thickness or the visibility of internal echogenic bands between children with adenoid hypertrophy and healthy controls.

H1 (Alternative Hypothesis): There is a difference in masseter muscle thickness or the visibility of internal echogenic bands between children with adenoid hypertrophy and healthy controls.

Sample Size Calculation No prior studies were identified comparing masseter muscle thickness between children with adenoid hypertrophy and healthy controls. The sample size was calculated using G*Power software. Assuming a medium effect size (0.6), an alpha level of 0.05, and a power of 0.80, the required total sample size was determined to be 72 participants.

Ultrasound Evaluation of the Masseter Muscle

Masseter muscle thickness and the visibility of internal echogenic bands will be assessed bilaterally at rest and during maximum clenching (intercuspal position). Evaluations will be performed with participants in the supine position. The ultrasound probe will be placed:

* Transversely: Parallel to the inferior mandibular border along a line connecting the oral commissure and the tragus.
* Longitudinally: Perpendicular to the mandibular body.

Thickness measurements (mm) will be taken from the thickest part of the muscle in both positions. Visibility of internal echogenic bands will be classified as follows:

* Type 1: Clear visibility of thin transverse bands.
* Type 2: Thickened bands with reduced echogenicity.
* Type 3: Disappearance or reduction in the number of bands.

Evaluations will be performed by the investigator (SY) at the Department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Aydın Adnan Menderes University.

Clinical Examination The principal investigator (BMA) will record each participant's age, sex, adenoid hypertrophy grade, occlusion type, molar relationship classification, overjet, overbite, number of carious, missing, and filled teeth, and the presence of mouth breathing and bruxism.

Statistical and Analytical Methods Data will be analyzed using SPSS version 19.0 (IBM Corp.). The Kolmogorov-Smirnov test will be used to assess normality of distribution. Categorical variables will be expressed as frequencies and percentages; continuous variables will be presented as means and standard deviations. The independent samples t-test will be used to compare measurement data between groups. The chi-square test will be used to evaluate associations between categorical variables and adenoid hypertrophy.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3 and 8 years
* Children diagnosed with adenoid hypertrophy
* Children without any systemic disease

Exclusion Criteria:

* Children with a history of surgery for adenoid hypertrophy
* Children who are uncooperative during clinical examination
* Children with syndromes involving the maxillofacial region
* Children with multiple missing teeth

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 3 to 8 years, with or without adenoid hypertrophy. The adenoid hypertrophy group will include pediatric patients diagnosed by the Department of Otorhinolaryngology at Aydın Adnan Menderes University Faculty of Medicine and scheduled for surgery. The control group will include healthy children without systemic disease who present to the Department of Pedodontics at Aydın Adnan Menderes University Faculty of Dentistry for routine dental examination.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Masseter Muscle Thickness and Internal Echogenic Bands Assessed by Ultrasonography | At enrollment (single assessment)
  The masseter muscles of both groups will be evaluated using a LOGIQ S8 R4 ultrasound device with a 9L linear probe. All participants will be examined in the supine position. The probe will be placed:
  Transversely: Along a line extending from the oral commissure to the ear tragus Longitudinally: Perpendicular to the mandibular body The thickness of the right and left masseter muscles will be measured in millimeters, both at rest and during maximum clenching, from the thickest region of the muscle.
  Internal echogenic bands will be classified into three types:
  * Type 1: Clear, thin transverse bands
  * Type 2: Thickened bands with reduced echogenicity
  * Type 3: Disappearance or reduction in the number of bands

SECONDARY OUTCOMES:
Primary Molar Occlusion (Mesial Step, Distal Step, Flush Terminal Plane) or Angle's Classification (Class I-III) of Permanent Molars in Children With and Without Adenoid Hypertrophy | At enrollment (single assessment)
  Evaluations will be conducted with children in maximum intercuspation. Primary molar occlusion (mesial step, distal step, flush terminal plane) will be recorded in children with primary dentition. Angle's classification (Class I-III) will be used in children with fully erupted permanent first molars.
  Primary occlusal classification will be based on the distal surfaces of the second primary molars. In a mesial step, the distal surface of the mandibular second primary molar is mesial to that of the maxillary molar. In a distal step, it is distal. In a flush terminal plane, the distal surfaces are aligned.
  Angle's classification will be recorded as follows: Class I, the mesiobuccal cusp of the mandibular first permanent molar aligns with the mesiobuccal groove of the maxillary molar; Class II, the cusp is distal to the groove; Class III, the cusp is mesial to the groove.
Overjet and Overbite in Children With and Without Adenoid Hypertrophy | At enrollment (single assessment)
  Participants will be seated in an upright position, with the head aligned parallel to the Frankfort horizontal plane. Measurements will be performed in maximum intercuspation.
  Overjet (Horizontal Measurement): The distance will be measured by drawing a perpendicular line from the incisal edge of the upper central incisor to the labial surface of the lower central incisor. A periodontal probe will be used, and the values will be recorded in millimeters (mm).
  Overbite (Vertical Measurement): The vertical distance between the incisal edges of the upper and lower central incisors will be measured along the labial surface of the lower incisor using a periodontal probe and recorded in millimeters (mm).
  If the upper or lower central incisors are missing or severely malpositioned, the measurements will be recorded as "not assessable."
Adenoid Hypertrophy Grade in Children Diagnosed With Adenoid Hypertrophy and Scheduled for Surgery | At enrollment (single assessment)
  The adenoid hypertrophy grade will be determined according to the degree of nasopharyngeal airway obstruction observed during otorhinolaryngological examination at Aydın Adnan Menderes University Faculty of Medicine, Department of Otorhinolaryngology, and will be classified into four grades. The participants with adenoid hypertrophy will consist of patients who were examined at the same department and scheduled for surgery. The degree of nasopharyngeal airway obstruction by the adenoid tissue will be assessed using endoscopic examination.
  Grade 1: Adenoid tissue occupies 0-25% of the nasopharyngeal airway; airway mostly patent, minimal or no obstruction.
  Grade 2: Occupies 26-50%; mild obstruction possible, nasal breathing generally intact.
  Grade 3: Occupies 51-75%; moderate obstruction, mouth breathing and snoring may occur.
  Grade 4: Occupies 76-100%; severe obstruction, marked mouth breathing, possible sleep-disordered breathing.
Presence of Mouth Breathing (Yes/No) in Children With and Without Adenoid Hypertrophy | At enrollment (single assessment)
  Mouth breathing will be assessed through both clinical observation and parental reporting. During clinical observation, children will be evaluated in an upright position at rest. The principal investigator will assess whether the child maintains lip closure and whether breathing occurs through the mouth. In addition, parents will be asked whether their child usually breathes through the mouth or nose during both wakefulness and sleep.
  Mouth breathing present (Yes): If the child breathes through the mouth at rest or if parents report that the child predominantly breathes through the mouth.
  Mouth breathing absent (No): If the child breathes through the nose at rest and parents do not report mouth breathing.
Number of Carious, Missing and Filled Teeth in Children With and Without Adenoid Hypertrophy | At enrollment (single assessment)
  The number of carious, missing, and filled teeth will be determined through clinical and radiographic examination.
Presence of Bruxism (Yes/No) in Children With and Without Adenoid Hypertrophy | At enrollment (single assessment)
  Bruxism will be assessed based on both parental reporting and clinical examination. Parents will be asked whether they have observed their child grinding or clenching their teeth during sleep or while awake. Clinical indicators such as abnormal tooth wear, masticatory muscle tenderness, and soft tissue signs (e.g., linea alba) will also be recorded to support the diagnosis.
  Bruxism present (Yes): If either parental report or clinical signs are observed.
  Bruxism absent (No): If neither parental reporting nor clinical signs are present.

CONTACTS AND LOCATIONS:
Overall Officials: Melis Akyıldız, phd, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Aydın Adnan Menderes University, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ariji Y, Sakuma S, Izumi M, Sasaki J, Kurita K, Ogi N, Nojiri M, Nakagawa M, Takenaka M, Katsuse S, Ariji E. Ultrasonographic features of the masseter muscle in female patients with temporomandibular disorder associated with myofascial pain. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Sep;98(3):337-41. doi: 10.1016/j.tripleo.2004.06.068. PMID 15356473